CLINICAL TRIAL: NCT05853718
Title: Study to Evaluate the Pharmacokinetic, Safety, and Efficacy of TAF in HBV-Infected Pregnant Women
Brief Title: Study of Tenofovir Alafenamide in HBV-Infected Pregnant Women
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-20210825-0020-01
Record Dates: First submitted 2023-04-26; First posted 2023-05-11 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Chronic Hepatitis b; Tenofovir Alafenamide Fumarate
Keywords: pharmacokinetics; CHB; TAF; pregnancy; mother-to-child transmission
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- TAF antiviral therapy group (Experimental): Eligible hepatitis B pregnant women are given TAF antiviral therapy (25mg, oral, 1/day) from week 28-32 of gestation until delivery
  Interventions: Drug: Tenofovir Alafenamide Tablets

INTERVENTIONS:
Drug: Tenofovir Alafenamide Tablets — Take 25mg TAF daily from week 28-32 of gestation until delivery
  Other Names: TAF

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, efficacy and safety of TAF in HBV-infected pregnant women.

DETAILED DESCRIPTION:
Pregnant women with high viral load (HBV DNA>2 × 10^5 IU/mL ) are recommended to be given Tenofovir Disoproxil Fumarate(TDF) for mother-to-child blocking of Chronic hepatitis B(CHB) by guidelines. Tenofovir alafenamide (TAF) is a new targeted pro-drug of Tenofovir (TFV) and was approved for use in China in December 2018. Compared with TDF, the therapeutic dose of TAF is small. 25mg TAF can obtain the antiviral effect similar to 300mg TDF, thus reducing the concentration of TFV in the blood.

This is a prospective clinical study, aiming to evaluate the pharmacokinetics, efficacy and safety of TAF in HBV-infected pregnant women when used for prevention of mother-to-child transmission of hepatitis B virus. 50 HBeAg-positive and HBV DNA levels ≥ 2 × 10^5 IU/mL pregnant women will be enrolled to receive Tenofovir alafenamide (TAF) from week 28-32 of gestation until delivery. According to the mother's wishes, intensive blood samples will be collected to determine the concentration of TAF and TFV in plasma of pregnant women before and after taking TAF, calculate the pharmacokinetic parameters. And the mother's milk is collected every day for 5 days for TAF concentration determination. The primary endpoint was the pharmacokinetic parameters of TAF and TFV, rate of mother-to-child transmission, the congenital malformation rate of infants. The secondary endpoint was the decrease of HBV DNA level at delivery, the clearance and seroconversion rate of HBeAg, postpartum ALT flare, concentration of TAF and TFV in milk,and other adverse events of mothers and infants.

ELIGIBILITY:
Inclusion Criteria:

* Age of 20-40 years; Positive for hepatitis B surface antigen (HBsAg) and hepatitis B virus e antigen (HBeAg); HBV DNA level >200 000 IU/mL during the 24th-32nd week of pregnancy; Willing to take TAF for mother-to-child blockade; Both husband and wife are willingly sign an informed consent.

Exclusion Criteria:

* Co-infected with hepatitis C or HIV, or other chronic diseases; History of spontaneous abortion or congenital malformation; Decompensated cirrhosis and liver cancer; History of kidney injury, CCr <50ml/min and urine protein test positive (>300mg/L); Fetal malformations detected by B-ultrasound during pregnancy; ALT > 2×upper limit of normal (ULN); TBIL ≥ 1×ULN; Albumin (ALB) < 25 g/L.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant woman is eligible for this study.
Enrollment: 50 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Assessment on the pharmacokinetics of TAF and TFV in plasma of pregnant women | The day before delivery
  When taking the last TAF before delivery , 2ml of drug-containing blood was collected from the upper extremity veins at 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24h after taking TAF. Blood drug concentration at each time point was calculated according to standard curve.
Rate of mother-to-child transmission of HBV | During 7-12 months after birth
  Testing for HBsAg in the infants between 7 and 12 months of age.
Rate of birth defect of infants | From the date of birth to age of 28 weeks
  The proportion of infants with the aforementioned abnormalities discovered during the study period

SECONDARY OUTCOMES:
Reduction of HBV DNA levels at delivery | At delivery
  Reduction of HBV DNA levels (IU/mL) at delivery when compared to the baseline before initiating TAF
Drug concentration of TAF and TFV in breast milk after drug withdrawal | Immediately after breast milk is available and last for 5 days
  Postpartum breast milk was collected to measure TAF and TFV concentrations after drug withdrawal
Concentrations of TAF and TFV in infant urine and plantar blood | Within 72 hours of birth
  Collect infant urine and plantar blood within 72 hours of birth

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyuan Ma, PhD, Principal Investigator — First People's Hospital of Hangzhou; Siying Li, MD, Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No